CLINICAL TRIAL: NCT05111535
Title: Stockholm Prospective Acute Kidney Injury Cohort Study
Brief Title: Stockholm Acute Kidney Injury Cohort
Acronym: SAKIS
Status: Completed | Type: Observational
Sponsor: Danderyd Hospital (Other)
Responsible Party: Principal Investigator, Jonas Spaak, Associate professor, Danderyd Hospital
Other Study IDs: SAKIS
Record Dates: First submitted 2021-09-24; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Acute Kidney Injury
Keywords: acute renal failure; hyperkalemia; major adverse cardiovascular event
MeSH Terms: conditions — Acute Kidney Injury; Hyperkalemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since 2009, adult patients with acute kindney injury (AKI) at the department of Nephrology, Danderyd University Hospital and Karolinska Institutet, have been included in a prospective cohort. All patients were treated and evaluated according to a detailed clinical memorandum, and data collected prospectively.

By 2020, 1861 patiens have been included of which 1519 fulfill current AKI criteria (as defined by KDIGO AKI guidelines) and will be evaluated regarding the following main research questions:

1. Descriptive study on patient characteristics, changes in biomarkers and in-hospital outcome.
2. One year outcome with focus on renal and cardiovascular outcomes.
3. Long-term outcome (up to 10 years) with focus on renal and cardiovascular outcomes.

DETAILED DESCRIPTION:
Acure kidney injury (AKI) remains a complex clinical challenge associated with high risk for short-term and long-term adverse events. Since 2009 patients with AKI at the department of Nephrology, Danderyd University Hospital and Karolinska Institutet, have been included in a prospective cohort. Adult patients with either s-creatinine >130 micromol/L and previously unknown level, or 30% increase from previous known level were included; patients on dialysis were not included. All patients were treated and evaluated according to a detailed clinical memorandum, and data collected prospectively.

By 2020, 1861 patiens have been included of which 1519 fulfill current AKI criteria and will be evaluated regarding the following main research questions:

1. Descriptive study on in-hospital outcome (death, renal recovery), patient characteristics, hyperkalemia and changes in biomarkers reflecting inflammation, acidosis and malnutrition.
2. One year outcome with focus on renal and cardiovascular outcomes (death, new dialysis, worsened renal function, myocardial infarction, stroke, or heart failure; MARCE).
3. Long-term outcome (up to 10 years) with focus on renal and cardiovascular outcomes (MARCE).

ELIGIBILITY:
Inclusion Criteria (one of the following):

* Serum creatinine (sCr) >130 µmol/l (1.47 mg/dl) at admission with previously unknown baseline,
* Increase in sCr by 30% from previous stable out-patient value.

Exclusion Criteria:

Ongoing dialysis treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective observational study, where all patients (aged 18 or above) with AKI admitted to the Department of nephrology at Danderyd University Hospital, Stockholm, Sweden, between 2009 and 2018 were included.
Sampling Method: Non-Probability Sample
Enrollment: 1861 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
In-hospital outcome | From admission until discharge or death, assessed for a period of up to 3 months
  Death
1-year outcome | From admission until 1 year
  Descriptive study on Major Adverse Renal or Cardiovascular Events (death, new dialysis, worsened renal function, myocardial infarction, stroke, or heart failure; MARCE)
Long-term outcome | From admission until 10 years
  Descriptive study on Major Adverse Renal or Cardiovascular Events (MARCE)

SECONDARY OUTCOMES:
In-hospital partial renal recovery | From admission until discharge or death, assessed for a period of up to 3 months
  Renal recovery by 30% at the time of discharge or death
In-hospital renal recovery | From admission until discharge or death, assessed for a period of up to 3 months
  Renal recovery by 50% at the time of discharge or death
In-hospital biomarkers | From previous values or values at admission until discharge or death, assessed for a period of up to 3 months
  Changes in biomarkers with focus on potassium, malnutrition, inflammation and acidosis

CONTACTS AND LOCATIONS:
Overall Officials: Christina Montgomerie, MD, Study Director — Karolinska Institutet and Danderyd University Hospital
Locations (2):
- Sweden (2):
  - Karolinska Institute at Danderyd University Hospital, Danderyd, Stockholm County
  - Danderyd University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided
Data may be shared, pending application and approval for the specific research question from the Swedish Ethical Review Authority